CLINICAL TRIAL: NCT00183053
Title: Trial of Proximity Alarms to Reduce Patient Falls
Brief Title: Proximity Alarms to Reduce Patient Falls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0050; R01AG025285 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Aging
Keywords: Hospitalization; Fall Risk; Frailty
MeSH Terms: conditions — Frailty

INTERVENTIONS:
Device: BedEx Patient Occupancy Monitoring System

SUMMARY:
The purpose of this study is to test an intervention to introduce and implement proximity alarms on the risk of falls in hospitalized patients.

DETAILED DESCRIPTION:
Proximity alarm systems are promoted as an approach to reduce falls and decrease use of physical restraints in hospitals, but they have not been tested rigorously. This study will implement proximity alarms at Methodist-University Hospital (M-UH), a 652-bed urban community hospital in Memphis, Tennessee. The hospital provides primary to tertiary care to a diverse adult patient population. The group randomized trial will be conducted on 16 25-bed general medical-surgical nursing units at M-UH. Nursing units will be randomized within blocks of 2 based on rates of falls that occur during an initial 3-month observation period. Over a 15-month intervention, 8 nursing units will be randomized to receive the alarm-based intervention, and 8 will utilize existing nursing care methods to minimize falls. Intervention units will receive an adequate supply of proximity alarm monitoring systems to apply to all patients considered by nursing staff to be at high risk for falls. An implementation team, consisting of a nurse-champion, geriatrician and biomedical instrumentation specialist, will train and conduct regular follow-up on intervention units to address technical issues related to use of the alarms. The primary outcome measure, patient falls, will be ascertained prospectively by a nurse-manager using a method developed to collect patient (e.g., orientation and postural blood pressure) and environmental data collected in a standardized manner. The primary aim of the study is to determine whether proximity alarm monitoring reduces falls. The study has been designed to test the hypothesis that patient falls will be 25% lower on intervention units compared to control units. The secondary aims are to determine whether proximity alarm monitoring reduces the use of physical restraints, or decreases patient care costs. This will be the first methodologically sound study to evaluate this promising approach to reducing falls in hospitals. Whether or not alarms successfully reduce falls, findings from this study have the potential to widely impact purchasing decisions and clinical practice related to fall prevention in acute-care settings.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to one of 16 study units at Methodist University Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Patient falls over 15 months

SECONDARY OUTCOMES:
Restraint use
patient care costs over 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald I. Shorr, MD, MS, Principal Investigator — Department of Aging & Geriatric Research, University of Florida
Locations (1):
- Methodist-University Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Tideiksaar R, Feiner CF, Maby J. Falls prevention: the efficacy of a bed alarm system in an acute-care setting. Mt Sinai J Med. 1993 Nov;60(6):522-7. PMID 8121429
- [Background] Morse JM. Enhancing the safety of hospitalization by reducing patient falls. Am J Infect Control. 2002 Oct;30(6):376-80. doi: 10.1067/mic.2002.125808. PMID 12360147
- [Background] Bates DW, Pruess K, Souney P, Platt R. Serious falls in hospitalized patients: correlates and resource utilization. Am J Med. 1995 Aug;99(2):137-43. doi: 10.1016/s0002-9343(99)80133-8. PMID 7625418
- [Background] Morse JM, Black C, Oberle K, Donahue P. A prospective study to identify the fall-prone patient. Soc Sci Med. 1989;28(1):81-6. doi: 10.1016/0277-9536(89)90309-2. PMID 2928815
- [Background] Oliver D, Britton M, Seed P, Martin FC, Hopper AH. Development and evaluation of evidence based risk assessment tool (STRATIFY) to predict which elderly inpatients will fall: case-control and cohort studies. BMJ. 1997 Oct 25;315(7115):1049-53. doi: 10.1136/bmj.315.7115.1049. PMID 9366729
- [Derived] Shorr RI, Chandler AM, Mion LC, Waters TM, Liu M, Daniels MJ, Kessler LA, Miller ST. Effects of an intervention to increase bed alarm use to prevent falls in hospitalized patients: a cluster randomized trial. Ann Intern Med. 2012 Nov 20;157(10):692-9. doi: 10.7326/0003-4819-157-10-201211200-00005. PMID 23165660